CLINICAL TRIAL: NCT06065410
Title: Research Assistant Doctor
Brief Title: The Effect of Intrinsic Focus on Gait Cycle and the Possible Confounding Effect of Noise in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Dilek Sayar, Research Assistant Medical Doctor, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Gazi University PMR.
Record Dates: First submitted 2023-08-08; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; white noise; intrinsic focusing; environmental sound
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: Between the ages of 50 and 75 years, who were admitted to the outpatient clinic of Gazi University Faculty of Medicine, Department of Physical Medicine and Rehabilitation or hospitalized in the ward and diagnosed with knee osteoarthritis according to ACR knee osteoarthritis criteria and had a Kellgren Lawrence staging of at least 2, were included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with knee osteoarthritis (Experimental)
  Interventions: Other: Baseline; Other: Intrinsic focus; Other: White noise; Other: environmental sound

INTERVENTIONS:
Other: Baseline — Walking without any instruction or sound
Other: Intrinsic focus — Walking focusing on ensuring equal step lengths and step durations on both sides and symmetry between both steps
Other: White noise — Intrinsic focus accompanied by white noise
Other: environmental sound — Intrinsic focus accompanied by environmental sound

SUMMARY:
Patients with knee osteoarthritis may develop an antalgic gait over time due to pain in the knee, characterized by a decrease in the stance phase and stride length on the painful side. Gait asymmetry, which may lead to different musculoskeletal problems in the future, is observed in the patients. Gait symmetry can be achieved with gait retraining, and effective focus is required during training.

In the literature, there are many studies of the positive effects of white noise on focusing, but there are also studies that report that it reduces focusing.

Today, exercise training is usually performed in rehabilitation units or on treadmills. As there are important differences between walking on a treadmill and walking outdoors in terms of noise, uneven ground and visual stimuli, the place where walking training is performed does not reflect the outdoor environment.

It was aimed to investigate the effect of internal focusing on gait cycle and the effect of white noise and environmental sound on internal focusing in patients with knee osteoarthritis

DETAILED DESCRIPTION:
A total of 40 patients between the ages of 50 and 75 years, who were admitted to the outpatient clinic of Gazi University Faculty of Medicine, Department of Physical Medicine and Rehabilitation or hospitalized in the ward and diagnosed with knee osteoarthritis according to ACR knee osteoarthritis criteria and had a Kellgren Lawrence staging of at least 2, were included.

The demographic data of the patients who were evaluated with the Hearing Handicap Inventory for the Elderly Screening Version (HHIE-S) and had adequate hearing level were recorded, bilateral true leg lengths were measured and detailed knee examinations were performed. Lequesne Knee Osteoarthritis Severity Index, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Lower Extremity Functional Scale (LEFS), 30 Second Sit to Stand Test and Timed Up and Go Test were applied to the patients who met the inclusion and exclusion criteria.

Patients walked at a speed of 0.40-0.45 m/s on a treadmill (Biodex Gait Trainer) where gait parameters were collected. Each patient walked at a constant speed for three minutes each in the baseline (without any instruction or sound), intrinsic focus (focusing on ensuring equal step lengths and step durations on both sides and symmetry between both steps), white noise (intrinsic focus accompanied by white noise) and environmental sound (intrinsic focus accompanied by environmental sound) conditions. After walking in each condition, gait parameters ( average step cycle, average step length, percentage of step length variability, percentage of left/right side stepping time and ambulation index) were recorded. The User Experience Questionnaire Short Form was adapted for our study to assess patients' experiences during intrinsically focused walking in white noise and environmental sound conditions. Patients were asked to rate their walking periods in white noise and environmental sound conditions in terms of inhibiting-supportive, inefficient-efficient, complex-simple, confusing-clear, boring-exciting, uninteresting-interesting, traditional-unique, and familiar-unusual characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Stable general condition
* Good cooperation
* Diagnosed with knee osteoarthritis according to ACR criteria
* At least stage 2 unilateral or bilateral knee osteoarthritis according to Kellgren Lawrence staging
* Individuals >50 years of age

Exclusion Criteria:

* Hearing Impairment Scale ≥ 26
* Presence of a neurological, cardiac or orthopedic pathology that prevents walking
* The presence of another pathology other than knee osteoarthritis that affects the knee and causes pain
* Presence of diseases such as osteoarthritis, gout, rheumatoid arthritis affecting other joints in the lower extremity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Average step cycle (cycle/second) | Evaluation at first visit of patients meeting the included criteria.12 minutes in total, with 3 minutes of assessment time in each walking condition
  After walking in each condition, average step cycle was recorded (total of 4 conditions)
Average step length (m) | Evaluation at first visit of patients meeting the included criteria.12 minutes in total, with 3 minutes of assessment time in each walking condition
  After walking in each condition, average step length was recorded (total of 4 conditions)
Percentage of step length variability (%) | Evaluation at first visit of patients meeting the included criteria. 12 minutes in total, with 3 minutes of assessment time in each walking condition
  After walking in each condition, percentage of step length variability was recorded (total of 4 conditions)
Percentage of left/right side stepping time (%) | Evaluation at first visit of patients meeting the included criteria.12 minutes in total, with 3 minutes of assessment time in each walking condition
  After walking in each condition, percentage of left/right side stepping time was recorded (total of 4 conditions)
Ambulation index | Evaluation at first visit of patients meeting the included criteria.12 minutes in total, with 3 minutes of assessment time in each walking condition
  After walking in each condition, ambulation index was recorded (total of 4 conditions)

SECONDARY OUTCOMES:
The User Experience Questionnaire Short Form | Evaluation was performed immediately after execution in white noise and environmentel sound conditions
  The User Experience Questionnaire Short Form was adapted for our study to assess patients' experiences during intrinsically focused walking in white noise and environmental sound conditions. Patients were asked to rate their walking periods in white noise and environmental sound conditions in terms of inhibiting-supportive, inefficient-efficient, complex-simple, confusing-clear, boring-exciting, uninteresting-interesting, traditional-unique, and familiar-unusual characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roos EM, Arden NK. Strategies for the prevention of knee osteoarthritis. Nat Rev Rheumatol. 2016 Feb;12(2):92-101. doi: 10.1038/nrrheum.2015.135. Epub 2015 Oct 6. PMID 26439406
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Turcot K, Armand S, Lubbeke A, Fritschy D, Hoffmeyer P, Suva D. Does knee alignment influence gait in patients with severe knee osteoarthritis? Clin Biomech (Bristol). 2013 Jan;28(1):34-9. doi: 10.1016/j.clinbiomech.2012.09.004. Epub 2012 Oct 12. PMID 23063098
- [Background] Neumann DL. A Systematic Review of Attentional Focus Strategies in Weightlifting. Front Sports Act Living. 2019 Aug 9;1:7. doi: 10.3389/fspor.2019.00007. eCollection 2019. PMID 33344931
- [Background] Johnson L, Burridge JH, Demain SH. Internal and external focus of attention during gait re-education: an observational study of physical therapist practice in stroke rehabilitation. Phys Ther. 2013 Jul;93(7):957-66. doi: 10.2522/ptj.20120300. Epub 2013 Apr 4. PMID 23559523
- [Background] Wulf G, Prinz W. Directing attention to movement effects enhances learning: a review. Psychon Bull Rev. 2001 Dec;8(4):648-60. doi: 10.3758/bf03196201. PMID 11848583
- [Background] Faisal AA, Selen LP, Wolpert DM. Noise in the nervous system. Nat Rev Neurosci. 2008 Apr;9(4):292-303. doi: 10.1038/nrn2258. PMID 18319728
- [Background] Muzet A. Environmental noise, sleep and health. Sleep Med Rev. 2007 Apr;11(2):135-42. doi: 10.1016/j.smrv.2006.09.001. Epub 2007 Feb 20. PMID 17317241
- [Background] Shidara M, Richmond BJ. Effect of visual noise on pattern recognition. Exp Brain Res. 2005 May;163(2):239-41. doi: 10.1007/s00221-005-2230-0. Epub 2005 Mar 15. PMID 15912370
- [Background] Helps SK, Bamford S, Sonuga-Barke EJ, Soderlund GB. Different effects of adding white noise on cognitive performance of sub-, normal and super-attentive school children. PLoS One. 2014 Nov 13;9(11):e112768. doi: 10.1371/journal.pone.0112768. eCollection 2014. PMID 25393410
- [Background] van Kempen E, van Kamp I, Lebret E, Lammers J, Emmen H, Stansfeld S. Neurobehavioral effects of transportation noise in primary schoolchildren: a cross-sectional study. Environ Health. 2010 Jun 1;9:25. doi: 10.1186/1476-069X-9-25. PMID 20515466